CLINICAL TRIAL: NCT05930873
Title: Evaluating the Effect of Immersive Room Intervention on Visual Attention in Children With Autism Spectrum Disorders
Brief Title: Immersive Room for Visual Attention in Children With Autism Spectrum Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Collaborators: Fondazione di Comunità Messina onlus (Unknown)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2023-002
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: autism; children; applied behavior analysis
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): treatment within an immersive room
  Interventions: Behavioral: Immersive room
- control group (Placebo Comparator): Traditional Treatment by presenting image stimuli in a paper format
  Interventions: Behavioral: stimuli in a paper format

INTERVENTIONS:
Behavioral: Immersive room — The intervention will be structured according to Applied Behavioral Analysis. A target stimulus will be presented on one of the four walls of the immersive room and a set of stimuli, including the target stimulus, which the subject will have to touch within a certain latency time.
  There will also be a hierarchy of prompts (least to most) in case the child gives an inaccurate answer or does not answer within the established time.
  Finally, as the last element of the behavioral chain, a social reinforcement will be delivered (a sound stimulus indicating applause) when the desired response is emitted.
  The intervention will be divided into phases, according to a progressive increase of the task in terms of visual attention, and an achievement of the acquisition criterion. Furthermore, each participant will be subjected to stimuli belonging to different semantic categories (fruit, animals, means of transport, clothing, figures and faces).
  Arms: experimental group
Behavioral: stimuli in a paper format — The intervention will be structured according to Applied Behavioral Analysis. A target stimulus will be presented in a paper format and a set of stimuli, including the target stimulus, which the subject will have to indicate within a certain latency time.
  There will also be a hierarchy of prompts (least to most) in case the child gives an inaccurate answer or does not answer within the established time.
  Finally, as the last element of the behavioral chain, a social reinforcement will be delivered (a sound stimulus indicating applause) when the desired response is emitted.
  The intervention will be divided into phases, according to a progressive increase of the task in terms of visual attention, and an achievement of the acquisition criterion. Furthermore, each participant will be subjected to stimuli belonging to different semantic categories (fruit, animals, means of transport, clothing, figures and faces).
  Arms: control group

SUMMARY:
Autism spectrum disorder (ASD) is a common neurodevelopmental disorder characterized by language delay, impaired social interactions, and repetitive behaviors. Its manifestation varies among individuals due to genetic and environmental factors. Technology-based interventions, such as robots, serious games, virtual reality and immersive room, have shown better results in the cognitive-behavioral treatment of ASD. Visual attention, which is often deficient in individuals with ASD, is a focus in these interventions, as it can aid stimulus processing. Virtual reality offers a more ecological environment for such interventions.

In this study, it has been demonstrated the effectiveness of virtual reality training by comparing the performance of an ASD group delivering treatment through the immersive room with a control group delivering traditional treatment.

Fifteen children with ASD between the ages of 5 and 10 years, with IQs between 55 and 85 will be included in the trial and, following an assessment related to visual attention processes, will be randomly assigned to the control group and the experimental group. The trial participants will, first, undergo structured sessions to foster or increase the receptive area related to the stimuli to which they will be subjected during the training.

ELIGIBILITY:
Inclusion Criteria:

* Child with diagnosis of autism

Exclusion Criteria:

* presence of other medical disorders

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) | The evaluation session will be scheduled pre-intervention. The test needs approximately 65-80 minutes to complete.
  Wechsler Intelligence Scale for Children Fourth edition (WISC-IV) is a clinical tool for assessing the cognitive abilities of children and young people between the ages of 6 years and 16 years and 11 months.
NEPSY-II | The evaluation sessions will be scheduled pre and post intervention.The test needs approximately 90 minutes to complete for preschool children and 120-180 minutes for school-age children
  NEPSY-II is the most internationally known battery for assessing neuropsychological development in developmental age.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 5th ed.; American Psychiatric Publishing: Washington, DC, USA, 2013.
- [Background] Zhang M, Ding H, Naumceska M, Zhang Y. Virtual Reality Technology as an Educational and Intervention Tool for Children with Autism Spectrum Disorder: Current Perspectives and Future Directions. Behav Sci (Basel). 2022 May 10;12(5):138. doi: 10.3390/bs12050138. PMID 35621435
- [Background] Nyaz Didehbani, Tandra Allen, Michelle Kandalaft, Daniel Krawczyk, Sandra Chapman,Virtual Reality Social Cognition Training for children with high functioning autism,Computers in Human Behavior,Volume 62, 2016,Pages 703-711
- [Background] McPartland JC, Webb SJ, Keehn B, Dawson G. Patterns of visual attention to faces and objects in autism spectrum disorder. J Autism Dev Disord. 2011 Feb;41(2):148-57. doi: 10.1007/s10803-010-1033-8. PMID 20499148
- [Background] Jiang, M., & Zhao, Q. (2017). Learning Visual Attention to Identify People with Autism Spectrum Disorder. In Proceedings - 2017 IEEE International Conference on Computer Vision, ICCV 2017 (pp. 3287-3296)
- [Background] Burgess PW, Alderman N, Forbes C, Costello A, Coates LM, Dawson DR, Anderson ND, Gilbert SJ, Dumontheil I, Channon S. The case for the development and use of "ecologically valid" measures of executive function in experimental and clinical neuropsychology. J Int Neuropsychol Soc. 2006 Mar;12(2):194-209. doi: 10.1017/S1355617706060310. PMID 16573854